CLINICAL TRIAL: NCT01038388
Title: A Phase I Trial Evaluating the Safety and Efficacy of Vorinostat (Zolinza ®) + RVD (Lenalidomide {Revlimid ®} + Bortezomib {Velcade ®} + Dexamethasone) for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: A Study of the Combination Vorinostat With Lenalidomide, Bortezomib and Dexamethasone for Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Jonathan Kaufman, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00017528; 1591 (Other: Other); RV-MM-PI-0420 (Other: Winship Cancer Institute)
Record Dates: First submitted 2009-07-07; First posted 2009-12-24 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib, lenalidomide, dexamethasone, vorinostat (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11; lenalidomide by mouth once a day on days 1-14; dexamethasone by mouth once a day on days 1, 2, 4, 5, 8, 9, 11, and 12; and vorinostat by mouth on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  After 8 courses, patients may receive maintenance therapy comprising lenalidomide by mouth once a day on days 1-21, dexamethasone by mouth once a day on days 1, 2, 8, and 9, and bortezomib IV over 3-5 seconds or subcutaneously on days 1 and 8. Courses may repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Vorinostat

INTERVENTIONS:
Drug: Bortezomib — 1.3mg/m² given IV or subcutaneously
  Other Names: Velcade
Drug: Lenalidomide — 25 mg given PO
  Other Names: Revlimid
Drug: Dexamethasone — 20 mg given PO
  Other Names: Decadron
Drug: Vorinostat — 100, 200, or 300 mg given PO
  Other Names: Zolinza

SUMMARY:
The purpose of the study is to evaluate the clinical effectiveness and side effects of the vorinostat, bortezomib, lenalidomide, and dexamethasone investigational combination.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the clinical effectiveness and side effects of the vorinostat, bortezomib, lenalidomide, and dexamethasone investigational combination.

All of these drugs - vorinostat, bortezomib, lenalidomide and dexamethasone, are approved by the FDA (U.S. Food and Drug Administration). They have not been approved in this combination for use in your type of cancer or any other type of cancer. Vorinostat is approved for treatment of patients with a different type of cancer (Cutaneous T-Cell Lymphoma). Bortezomib is currently approved for the treatment of multiple myeloma. Lenalidomide is currently approved for the treatment of certain types of myelodysplastic syndrome (another form of cancer affecting the blood) and for use with dexamethasone for patients with multiple myeloma who have received at least one prior therapy. Dexamethasone is commonly used, either alone, or in combination with other drugs, to treat multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma Diagnosis: Subject was previously diagnosed with multiple myeloma based on standard diagnostic criteria or by the new International Myeloma Foundation 2003 Diagnostic Criteria (ALL 3 REQUIRED):

  1. Monoclonal plasma cells in the bone marrow > 10% and/or presence of a biopsy-proven plasmacytoma.
  2. Monoclonal protein present in the serum and/or urine.
  3. Myeloma-related organ dysfunction (1 or more).

     * [C] Calcium elevation in the blood S. Calcium >10.5 mg/l or upper limit of normal{}.
     * [R] Renal insufficiency S. Creatinine > 2 mg/dl{}.
     * [A] Anemia Hemoglobin < 10 g/dl or 2 g < normal{}.
     * [B] Lytic bone lesions or osteoporosis.
* Patient must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma.

  * Prior treatment of hypercalcemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period).
  * Bisphosphonates are permitted
* Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible. One week must have lapsed since last date of radiotherapy, which is recommended to be a limited field. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and one week have passed since the last date of therapy.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-international unit (mIU)/mL 10 - 14 days prior to therapy and repeated again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Age ≥ 18 years at the time of signing Informed Consent.
* All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrollment.
* Subject has a Karnofsky performance status of ≥ 60.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Patient has ≥ Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment.
* Renal insufficiency (serum creatinine levels > 2.5 mg/dL).
* Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count ≥ 50,000 cells/mm³).
* Subjects with an absolute neutrophil count (ANC) < 1000 cells/mm³. Growth factors may not be used to meet ANC eligibility criteria.
* Subjects with a hemoglobin < 8.0 g/dL.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN).
* Concomitant therapy medications that include corticosteroids (except as indicated in inclusion criteria).
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Clinically relevant active infection requiring intravenous antibiotics.
* Serious co-morbid medical conditions such as chronic obstructive or chronic restrictive pulmonary disease, and cirrhosis.
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
* Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or if the expected survival from other malignancy is greater than 90% at 5 years.
* Female subject is pregnant or breast-feeding.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Uncontrolled diabetes mellitus (Fasting Blood Sugar > 400 despite medical treatment).
* Hypersensitivity to acyclovir or similar anti-viral drug.
* Known history of POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
* Known HIV infection .
* Known active hepatitis B or C viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended phase II doses (RP2D) of vorinostat in combination with lenalidomide, bortezomib, and dexamethasone. | Every 3 weeks

SECONDARY OUTCOMES:
Efficacy by standard myeloma measurements (SPEP, UPEP [urine protein electrophoresis], bone marrow) | Every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kaufman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States